CLINICAL TRIAL: NCT04543071
Title: A Phase 2 Study With Combination Chemotherapy (Gemcitabine and Nab-Paclitaxel), Chemokine (C-X-C) Motif Receptor 4 Inhibitor (BL-8040), and Immune Checkpoint Blockade (Cemiplimab) in METastatic Treatment naïve PANCreas Adenocarcinoma
Brief Title: Chemo4METPANC Combination Chemokine Inhibitor, Immunotherapy, and Chemotherapy in Pancreatic Adenocarcinoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Gulam Manji (Other)
Collaborators: Regeneron Pharmaceuticals (Industry); BioLine Rx (Unknown)
Responsible Party: Sponsor-Investigator, Gulam Manji, Assistant Professor of Medicine, Columbia University
Organization: Columbia University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AAAS9513
Record Dates: First submitted 2020-08-10; First posted 2020-09-09 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: Pancreatic Cancer; Adenocarcinoma of the Pancreas; Adenocarcinoma
MeSH Terms: conditions — Pancreatic Neoplasms; Adenocarcinoma | interventions — 4-fluorobenzoyl-TN-14003; cemiplimab; Gemcitabine; Taxes; Albumin-Bound Paclitaxel

STUDY DESIGN:
Intervention Model Description: The study will use a Simon optimal 2-stage design. The study will enroll 10 participants in the first stage. If 3 or more participants meet the endpoint in the first stage, the study will be expanded to a total of 40 participants. If a total of 14 or more participants achieve CR or PR by 16 weeks weeks, the agents will warrant further study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Motixafortide, Cemiplimab, Gemcitabine, Nab-Paclitaxel (Experimental): Participants will receive standard FDA-approved doses of gemcitabine and nab-paclitaxel for pancreas cancer and cemiplimab at the dose that is approved for participants with skin cancer. Participants will also receive motixafortide at a dose that has been deemed safe in previous studies when used in combination with immunotherapy and chemotherapy. If the combination study treatment causes a serious side effect in participants, the study treatment will be modified.
  Interventions: Drug: Motixafortide; Drug: Cemiplimab; Drug: Gemcitabine; Drug: Nab paclitaxel

INTERVENTIONS:
Drug: Motixafortide — 1.25 mg/kg subcutaneous (SC) monotherapy daily for 5 days during priming, followed by twice weekly
  Other Names: BL-8040
Drug: Cemiplimab — 350 mg intravenous (IV) once every 21 days
  Other Names: REGN2810
Drug: Gemcitabine — 1000 mg/m2 IV on days days 1, 8, 14 (every 28 days)
  Other Names: Gemzar
Drug: Nab paclitaxel — 125 mg/m2 IV on days 1, 8, 14 (every 28 days)
  Other Names: Abraxane

SUMMARY:
The purpose of this study is to determine if combination treatment with cemiplimab, motixafortide, gemcitabine, and nab-paclitaxel is effective in decreasing the size of the tumor(s), if it will prolong life in patients, and if it's safe. The treatment consists of standard chemotherapy (gemcitabine and nab-paclitaxel) which is FDA approved and is standard treatment for patients with pancreatic adenocarcinoma. Participants will receive immunotherapy (cemiplimab) which activates the body's immune system to attack cancer cells. Cemiplimab is FDA approved for treatment of skin cancer but not for pancreas cancer. Participants will also receive Motixafortide, a new medication which has shown in the laboratory to help immunotherapy work better. Motixafortide has been tested together with immunotherapy (Pembrolizumab), and chemotherapy (5-Fluorouracil and liposomal Irinotecan) and was deemed safe to test additional patients. Motixafortide has not been tested with the specific immunotherapy (Cemiplimab) and chemotherapy (gemcitabine and nab-paclitaxel) which participants will receive and is being tested in this clinical trial.

DETAILED DESCRIPTION:
Pancreas adenocarcinoma (PDAC) is an aggressive pancreatic cancer for which little progress has been made towards effective treatment. This is a Phase 2 open-label, multi-center study for patients with treatment-naïve metastatic PDAC. The goal of the study is to assess the preliminary efficacy of a CXCR4 antagonist (motixafortide), (cemiplimab), gemcitabine and nab-paclitaxel compared based on the response rate to historical controls in first line metastatic PDAC. Subjects will be treated with 5 days of motixafortide daily alone in the priming phase, followed by motixafortide twice a week, cemiplimab once every three weeks and and standard of care chemotherapy (gemcitabine and nabpaclitaxel).

ELIGIBILITY:
Inclusion criteria:

1. Histological or pathological confirmation of metastatic pancreas adenocarcinoma

   1. Cytologic or histologic proof of pancreas adenocarcinoma needs to be verified by the treating institution pathologist, either from the initial diagnostic biopsy or from the required pre-treatment biopsy, prior to initiation of any study-related therapy.
   2. Pathologic confirmation of metastatic (stage IV) disease (unresectable) on research pretreatment biopsy is required prior to initiation of therapy.
   3. Patients with endocrine or acinar pancreatic carcinoma are not eligible for the study.
2. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
3. Age ≥18 years
4. Adequate hematological and end-organ function (test results from within 14 days prior to initiation of study treatment):

   1. Absolute Neutrophil Count (ANC) ≥ 1.5 x 109/L without granulocyte colony-stimulating factor support
   2. White Blood Cell Count (WBC) count ≥ 2.5 x 109 /L (2500/uL)
   3. Lymphocyte count ≥ 0.5 x 109/L (500/uL)
   4. Platelet count ≥ 100 x 109/L (100,000/uL) without transfusion
   5. Hgb ≥ 9.0 g/dL
   6. Aspartate aminotransferase (AST), alanine transaminase (ALT), and alkaline phosphatase (ALP) ≤ 2.5X upper limit of normal (ULN), unless elevated secondary to biliary obstruction from the pancreas mass and amenable to decompression prior to initiation of therapy
   7. Serum total bilirubin ≤ 1.5X ULN, unless in patients with known Gilbert disease (≤ 3X ULN), or unless elevated secondary to biliary obstruction from the pancreas mass and amenable to decompression prior to administration of investigational therapy
   8. Albumin ≥ 3.5 g/dL
   9. Creatinine within ULN or calculated creatinine clearance (CrCl) >50 mL/min using the Cockcroft-Gault formula
   10. International normalized ratio (INR) and activated partial thromboplastin time (aPTT) ≤ 1.5X ULN, except for those on stable anticoagulation for at least two weeks
5. Measurable disease according to Immune Modified (IM)-RECIST and tumor accessible for fresh biopsy
6. Negative pregnancy test: Women of child-bearing potential must have a negative serum pregnancy test at screening and must agree to use an effective form of contraception from the time of the negative pregnancy test until a minimum of 3 months after the last dose of study drug. Effective forms of contraception include abstinence, hormonal contraceptive (injectable or implantable) in conjunction with a barrier method. Women of non-child-bearing potential must have been postmenopausal for ≥ 1 year or surgically sterile.
7. Birth control agreement: Fertile men must agree to use an effective method of birth control with female partners of childbearing potential (condoms plus an additional contraceptive method such as an injectable or implantable hormonal contraceptive) during the study and for up to 3 months after the last dose of study drug.
8. Informed consent: Participants must be willing and able to provide written informed consent prior to any study-related procedures and to comply with all study requirements.
9. Ability to comply: Participants must be able to comply with the study protocol, according to the investigator's judgement.
10. DVT testing Participants must have undergone lower extremity dopplers to rule out deep venous thrombosis (DVT) within the screening period, and undergo therapeutic anticoagulation if evidence of DVT is identified.
11. Anticoagulation treatment Subjects who are stable on full-dose anticoagulation medication for at least 2 weeks are considered eligible. However, subjects who have an increased clot burden on full-dose anticoagulation, such as central pulmonary embolism, or peripheral pulmonary embolism, and DVT within the extremities will be considered eligible only with the approval of the Principal Investigator.

Exclusion criteria:

1. Prior systemic therapy for PDAC: Participants may not have had systemic chemotherapy, investigational therapy, or treatment with T-cell co-stimulating or immune check point blockade therapies (including anti-CTLA-4, anti PD-1, and anti PD-L1 therapeutic antibodies) prior to initiation of study treatment.
2. Prior radiation therapy for PDAC Participants may not have had radiation therapy to within two weeks prior to initiation of study treatment. Participants may not have had previous radiotherapy to the primary pancreas lesion or a metastatic site except for palliation for pain. Participants who receive radiation to 25% or more of the bone marrow will be excluded.
3. Prior surgery for PDAC Participants may not have had surgical resection of PDAC prior to initiation of study treatment
4. Patients currently receiving any other investigational agents
5. Adverse events from prior anti-cancer therapy that have not resolved to Grade ≤ 1 or better, with the exception of alopecia of any grade and Grade ≤ 2 peripheral neuropathy
6. Concomitant treatment with other anti-neoplastic agents (hormone therapy acceptable)
7. Uncontrolled pleural effusion, pericardial effusion, or ascites. Subjects who required drainage within the four weeks prior or require pleural, pericardial, or peritoneal catheters for drainage are ineligible.
8. Uncontrolled tumor-related pain Patients requiring narcotic pain medication must be on a stable regimen for at least two weeks prior to study entry.
9. History of leptomeningeal or brain/ Central Nervous System (CNS) metastases
10. Uncontrolled hypercalcemia (ionized calcium > 1.5 mmol/L, calcium > 12 mg/dL, or corrected serum calcium > upper limit of normal) or symptomatic hypercalcemia requiring continued use of bisphosphonate therapy.
11. Recent major surgery or significant traumatic injury Participants may not have undergone major surgery or experienced significant traumatic injury within 14 days prior to initiating study treatment, or be recovering from procedure related adverse events of > Grade 1.
12. Active or history of autoimmune disease or immune deficiency Includes, but is not limited to, myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, antiphospholipid antibody syndrome, Wegener granulomatosis, Sjögren's syndrome, Guillain-Barré syndrome, or multiple sclerosis, with the following exceptions:

    1. Patients with a history of autoimmune-related hypothyroidism who are on stable thyroid-replacement hormone for the past three months are eligible for the study.
    2. Patients with controlled Type 1 diabetes mellitus who are on a stable insulin regimen for the past month are eligible for the study.
    3. Patients with eczema, psoriasis, lichen simplex chronicus, or vitiligo with dermatologic manifestations only (e.g., patients with psoriatic arthritis are excluded) are eligible for the study provided all of following conditions are met:

       * Rash must cover <10% of body surface area;
       * Disease is well-controlled at baseline and requires only low-potency topical corticosteroids;
       * No occurrence of acute exacerbations of the underlying condition requiring psoralen plus ultraviolet A radiation, methotrexate, retinoids, biologic agents, oral calcineurin inhibitors, or high-potency or oral corticosteroids within the previous 12 months.
13. History of idiopathic pulmonary fibrosis, interstitial lung disease, organizing pneumonia (e.g., bronchiolitis obliterans), drug-induced pneumonitis, or idiopathic pneumonitis, or evidence of active pneumonitis on screening chest computed tomography scan (history of radiation pneumonitis or fibrosis in the radiation field is permitted).
14. Positive for HIV at screening or any time prior to screening Patients without prior positive HIV test result will undergo an HIV test at screening, unless not permitted under local regulations.
15. Hepatitis B virus (HBV) infection (chronic or acute) Defined as having a positive hepatitis B surface antigen (HBsAg) test at screening. Patients with a past or resolved HBV infection, defined as having a negative HBsAg test and a positive total hepatitis B core antibody test at screening, are eligible for the study.
16. Active hepatitis C virus (HCV) infection: Defined as positive HCV antibody test followed by a positive HCV RNA test at screening.

    The HCV RNA test will be performed only for patients who have a positive HCV antibody test.
17. Known clinically significant liver disease, including alcoholic hepatitis, cirrhosis, fatty liver disease, and inherited liver disease.
18. Active tuberculosis
19. Infection: Patients may not have had a severe infection requiring antibiotic treatment within the two weeks prior to initiation of study treatment. This includes, but is not limited to, hospitalization for complications of infection, bacteremia, or severe pneumonia. However, patients who were admitted for biliary tract infection due to bile duct obstruction at time of diagnosis must have a functioning biliary stent (as evidenced by declining total bilirubin and ≤ 2X ULN) and resolved infection (defined by normalization of elevated white blood cell count, absence of signs of infection) and completion of an antibiotic course (at least a seven-day course) prior to initiation of therapy. Patients receiving prophylactic antibiotics (e.g., to prevent a urinary tract infection or chronic obstructive pulmonary disease exacerbation) are eligible for the study.
20. Significant cardiovascular disease: Patient may not have significant cardiovascular disease (such as New York Heart Association Class II or greater cardiac disease, myocardial infarction, or cerebrovascular accident) within 12 months prior to initiation of study treatment, seizure disorder, uncontrolled hypertension, or unstable arrhythmia or unstable angina within 3 months prior to initiation of study treatment.
21. Left ventricular ejection fraction below institutional lower limit of normal or below 50%, whichever is lower.
22. Baseline QTcF ≥ 450 ms (males) or ≥ 470 ms (females)
23. Grade ≥ 3 hemorrhage or bleeding event within 28 days prior to initiation of study treatment
24. Prior autologous stem cell, allogeneic stem cell, or solid organ transplantation
25. History of other malignancy Patient may not have a history of malignancy other than PDAC within two years prior to screening, with the exception of those with a negligible risk of metastasis or death (e.g., 5- year overall survival of > 90%), such as adequately treated carcinoma in situ of the cervix, non-melanoma skin carcinoma, localized prostate cancer, ductal carcinoma in situ, or Stage I uterine cancer.
26. Recent vaccination: Patients may not have been treated with a live, attenuated vaccine within four weeks prior to initiation of study treatment, or anticipate the need for such a vaccine during treatment with cemiplimab or within five months after the last dose of cemiplimab.
27. History of severe allergic anaphylactic reactions to chimeric or humanized antibodies or fusion proteins
28. Known allergy or hypersensitivity to any of the study drug excipients
29. Recent immunosuppressive treatment: Patients may not have been treated with systemic immunosuppressive medication (including, but not limited to, corticosteroids, cyclophosphamide, azathioprine, methotrexate, thalidomide, calcineurin inhibitors, and anti-tumor necrosis factor alpha agents) within two weeks prior to initiation of study treatment, or anticipate the need for systemic immunosuppressive medication during the course of the study, with the following exceptions:

    a. Patients who received a one-time pulse dose of systemic immunosuppressant medication are eligible for the study after approval from the Principal Investigator.
30. Pregnancy: Pregnant women are excluded from this study because there is an unknown, but potential risk for adverse events to the fetus. Breastfeeding should be discontinued prior to start of treatment because there is an unknown, but potential risk for adverse events in nursing infants secondary to treatment.
31. Other contraindicated conditions Any other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding that contraindicates the use of an investigational drug, may affect the interpretation of the results, or may render the patient at high risk from treatment complications in the opinion of the treating investigator.
32. Uncontrolled psoriasis, porphyria, proximal myopathy or neuropathy
33. Severe depression Subjects hospitalized for depression within the past two years, or who have prior suicidal attempts will be excluded.
34. Has received transfusions of blood products (including platelets or red blood cells) within 4 weeks prior to study Day 1.
35. Patients who received mineralocorticoids (e.g., fludrocortisone), corticosteroids for chronic obstructive pulmonary disease or asthma, or low-dose corticosteroids for orthostatic hypotension or adrenal insufficiency are eligible for the study if receiving equivalent to ≤ 10 mg of prednisone daily (10mg prednisone is equivalent to either cortisone - 50mg; hydrocortisone - 40mg; triamcinolone - 8mg; prednisolone - 10mg; methylprednisolone - 8mg; betamethasone - 1.5mg; or dexamethasone - 1.5mg). Patients receiving > 10 mg of prednisone or equivalent per day for greater than five days within 28 days of starting study related therapy are not eligible. Steroids administered prior to gemcitabine and nab-paclitaxel should be administered as per standard institutional guidelines.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2020-11-09 (Actual); Primary Completion 2028-06 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate (Complete Response (CR) + Partial Response (PR)) | 16 weeks
  Complete response is defined as the disappearance of all lesions. Partial response is defined as ≥30% decrease in the sum of diameters of target lesions, in the absence of CR, new lesions, and unequivocal progression in non-target lesions.

SECONDARY OUTCOMES:
Incidence of Treatment Related Toxicities | Up to 5 years
  All participants will be evaluable for toxicity from the time of their first treatment with the study drugs. The counts of treatment-related toxicities will be reported by type and severity according to the National Cancer Institute Common Terminology Criteria for Adverse Events, version 5.
Median Overall Survival | Up to 5 years
  Overall survival is defined as the time from the date of first treatment with study drug to the time of death from any cause or last follow-up if alive.
Median Progression Free Survival | Up to 5 years
  Progression free survival is defined as the time from first treatment with the study drug to the earliest of either disease progression or death from any cause.
Duration of Clinical Benefit | Up to 5 years
  Duration of clinical benefit is defined as the time from first treatment with the study drug to the earliest of either disease progression or death from any cause in subjects who achieved a CR, PR, or stable disease (SD).
Disease Control Rate | 16 weeks
  The number of participants that achieve disease control rate (CR+PR+SD) by 16 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Gulam Manji, MD,PhD, Principal Investigator — Columbia University
Locations (3):
- United States (3):
  - Columbia University Irving Medical Center, New York, New York
  - Brown University, Providence, Rhode Island
  - Medical College of Wisconsin, Wisconsin Diagnostic Labratories, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: Undecided